CLINICAL TRIAL: NCT00983411
Title: Impact of Non-intentional Leaks on Breathing Pattern and Work of Breathing During Non-invasive Ventilation: Study in Awakened Healthy Subjects and Awakened Obesity Hypoventilation Syndrome(OHS)Patients and During the Sleep in OHS Patients.
Brief Title: Impact of Non-intentional Leaks on Noninvasive Ventilation
Acronym: NIV-Leaks
Status: Completed | Type: Observational
Sponsor: AGIR à Dom (Other)
Responsible Party: Sponsor
Other Study IDs: AGIR-02
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2009-09

CONDITIONS: Intermittent Positive-pressure Ventilation; Respiratory Physiological Phenomena
Keywords: non-invasive intermittent positive-pressure ventilation; work of breathing; Pulse transit time

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy and OHS subjects: 10 healthy subjects: 20 to 60 years old 10 patients with Obesity hypoventilation syndrome: 20 to 70 years old treated with nocturnal non invasive ventilation for at least three months.
  Interventions: Other: Non intentional leaks during non invasive ventilation

INTERVENTIONS:
Other: Non intentional leaks during non invasive ventilation — During NIV sessions (in awake state for both the 10 healthy and the 10 OHS subjects and during sleep only for the OHS subjects), the investigators will create several levels of non intentional leaks in a random order

SUMMARY:
The investigators hypothesized that increasing non intentional leaks could increase work of breathing and could lead to patient/non-invasive ventilation (NIV) asynchrony.

The main objective is to compare ventilatory pattern (work of breathing, flow, pressure) under NIV with and without non-intentional leaks in 10 awakened healthy subjects and 10 awakened and asleep obese hypoventilation syndrome (OHS) patients.

Methods: While the subjects will be under NIV, several levels of leaks will be simulated in a random order with an automatically opening valve. Breathing pattern (work of breathing,flow, pressure, thorax and abdominal movements) will be recorded by Polygraphy. Healthy subjects will be recorded only during awakened state. OHS patients will be recorded both during awake and sleep sates.

Analysis: A repeated measures analysis of variance (ANOVA) will compare work of breathing according to the different levels of leaks.

ELIGIBILITY:
Inclusion Criteria:

* OHS patients, in stable stade, teated with nocturnal non invasive ventilation for at least three months.
* Healthy subjects without known pathology

Exclusion Criteria:

* OHS patients: instable cardio-respiratory status and/or acute cardio-respiratory failure three month before the inclusion. Latex allergy, oesophageal varices.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 healthy subjects recruited in professionnal area 10 patients with Obesity hypoventilation syndrome addressed to the sleep laboratory for clinical assessment
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Main outcome measure:Work of breathing assessed by measurement of oesophageal pressure according to the levels of non intentional leaks during non invasive ventilation | Oesophageal pressure will be assessed during all the duration of the study (2hours for the healthy subjects, overnight for the OHS patients)

SECONDARY OUTCOMES:
Secondary outcome measure: Assessments of the pulse transit time (PTT) and measurement of the oral opening (JAWSENS-NOMICS)according to the levels of non intentional leaks during non invasive ventilation | PTT and oral opening will be assessed during all the duration of the study (2hours for the healthy subjects, overnight for the OHS patients)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis Pepin, Pr, Principal Investigator — Laboratoire EFCR et Sommeil, CHU Grenoble
Locations (1):
- Laboratoire EFCR et Sommeil CHU Grenoble, Grenoble, France

REFERENCES:
- [Derived] Contal O, Carnevale C, Borel JC, Sabil A, Tamisier R, Levy P, Janssens JP, Pepin JL. Pulse transit time as a measure of respiratory effort under noninvasive ventilation. Eur Respir J. 2013 Feb;41(2):346-53. doi: 10.1183/09031936.00193911. Epub 2012 Apr 20. PMID 22523360